CLINICAL TRIAL: NCT05042648
Title: Role of Preoperative Transdermal Buprenorphine Patch in Reducing Postoperative Opioids Consumption in Patients Undergoing Total Knee Arthroplasties - A Randomised Controlled Trial.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Security Forces Hospital (Other)
Responsible Party: Principal Investigator, Anwar ul Huda, Consultant, Security Forces Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SecurityFH
Record Dates: First submitted 2021-09-04; First posted 2021-09-13 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-04

CONDITIONS: Patients Aged Between 18 and 65years Undergoing Total Knee Arthroplasty

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Group A) (No Intervention): Group A will receive no intervention
- Buprenorphine group (Group B) (Experimental): Group B will receive buprenorphine patch of 10 mg (sustained release of 10 µg/h) applied either on chest or on outer side of arm 12 h before surgery. The transdermal buprenorphine patch should be applied to intact skin on the flat surfaces of the upper outer arm, upper chest, upper back, or the side of the chest.
  Interventions: Drug: Buprenorphine patch

INTERVENTIONS:
Drug: Buprenorphine patch — Group B will receive buprenorphine patch of 10 mg (sustained release of 10 µg/h) applied either on chest or on outer side of arm 12 h before surgery. The transdermal buprenorphine patch should be applied to intact skin on the flat surfaces of the upper outer arm, upper chest, upper back, or the side of the chest. The skin should be dry, clean, non irritated, non hairy (hair should be trimmed with scissors, not shaved), and without large scars.
  Arms: Buprenorphine group (Group B)

SUMMARY:
This study will help us in understanding the role of transdermal buprenorphine patch in reducing consumption of opioids in patients undergoing total knee replacement. The objective of our study is to investigate the role of preoperative TDB patch in reducing postoperative opioids consumption in patients undergoing total knee arthroplasties. Patients aged between 18 and 65years, scheduled to undergo total knee arthroplasty with an ASA score of 1 to 3 will be included in the study.

DETAILED DESCRIPTION:
Effective postoperative pain control is a major challenge to the treating surgeons and Anaesthetists. Most opioids cause side effects such as sedation, nausea, vomiting, and respiratory depression. A number of other modalities have also been recommended for treatment of post-operative pain, including epidural infusion, patient-controlled analgesia, peripheral nerve block, continuous intra-articular infusion and local intra-articular analgesic injection. However, all of these treatments are invasive and aggressive and are potentially associated with regional bleeding, infection and nerve damage.

In the study by Londhe et al, all patients received peri-articular local anesthetic infiltration and then epidural/femoral nerve block infusion for 72 hours postoperatively. Group A received the TDB patch 5 mcg applied at the end of surgery. Group B received a combination of paracetamol and tramadol. They concluded that TDB patch is more efficacious in reducing postoperative pain after TKA surgery and can be safely used with fewer systemic side effects when compared to conventional analgesics.

The objective of our study is to investigate the role of preoperative TDB patch in reducing postoperative opioids consumption in patients undergoing total knee arthroplasties.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 65years, scheduled to undergo total knee arthroplasty with an ASA score of 1 to 3 will be included in the study.

Exclusion Criteria:

* Patients who will refuse enrollment or later request removal from the study, those who are unable to give informed consent and patients with contraindications for regional anesthesia like known allergy to local anesthetics, bleeding diathesis, use of anticoagulants or corticosteroids, inability to operate patient controlled analgesia (PCA) system, psychiatric disorders or use of psychiatric medications and known allergy to TDB patch.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-12-15 (Estimated); Study Completion 2023-12-15 (Estimated)

PRIMARY OUTCOMES:
morphine (PCA) consumption | 24 hours
  24 hours morphine consumption

SECONDARY OUTCOMES:
Pain score measured by Numeric rating scale (NRS) | 15th minute, 30th minute and 1st, 2nd, 6th, 12th, 18th and 24th hours
  NRS pain score at 15th minute, 30th minute and 1st, 2nd, 6th, 12th, 18th and 24th hours both at rest and on movement
Rescue analgesic use | 24 hours
  rescue analgesic use within the ﬁrst 24h.

OTHER OUTCOMES:
Postoperative nausea and vomiting | First 24 hours
  The severity of both nausea and sedation will be assessed by patients on a 4 point scale (none, mild, moderate, and severe). Nurses will note any vomiting in the recovery room or on the ward
Patient satisfaction | 24 hours
  patient satisfaction score will also be measured on score of 1-10.
range of motion (ROM) | 24 hours
  The range of motion (ROM) will be measured by the same physical therapist using a goniometer pre-operatively and on PD 1

CONTACTS AND LOCATIONS:
Locations (1):
- Security Forces Hospital Program, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
It will be shared on request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 2 years
Access Criteria: On request